CLINICAL TRIAL: NCT06124872
Title: Mapping Snakebite Risk in Kenya and Eswatini: Using Primary Data Collection and Geostatistical Techniques to Develop an Approach to Remote Risk Estimation for Snakebite
Brief Title: Mapping Snakebite Risk in Kenya and Eswatini
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); Institute of Primate Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: 22_060
Record Dates: First submitted 2023-05-03; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Snakebite; Epidemiology
MeSH Terms: conditions — Snake Bites | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Community survey 1 (planned demographic/health survey): Households included in a planned demographic and health survey (DSS).
  All participants included in this survey will be invited to respond to snakebite questions.
  Interventions: Other: Survey questionnaire
- Community survey 2 (Stand alone survey): 25 households randomly selected for inclusion within each survey cluster.
  Survey clusters will be randomly selected enumeration units within study Counties.
  Interventions: Other: Survey questionnaire
- Community survey 3 (Stand alone survey): 25 households randomly selected for inclusion within each survey cluster.
  Survey clusters will be randomly selected enumeration units within study Counties.
  Interventions: Other: Survey questionnaire
- Key informant interviews: Stakeholders in the process of healthcare decision making and research relevant to snakebite and snakebite envenoming
  Interventions: Other: Key informant interview

INTERVENTIONS:
Other: Survey questionnaire — Household screening questionnaire Snakebite details questionnaire where a history of snakebite is reported
  Groups: Community survey 1 (planned demographic/health survey); Community survey 2 (Stand alone survey); Community survey 3 (Stand alone survey)
Other: Key informant interview — Semi-structured interview with selected key informants
  Groups: Key informant interviews

SUMMARY:
The goal of this observational study is to learn about how snakebite risk varies in different environments in Kenya and understand how this information can be used to support decision makers.

The main questions it aims to answer are:

1. To what extent can information on snakebite cases and data on geographic, climatic and sociodemographic factors be used to predict geographical variation in snakebite risk in Kenya and Eswatini?
2. What is the most effective means of presenting outputs from spatial analysis of snakebite risk to ensure its effective use in research and healthcare decision making?

Participants in the community survey will be asked survey questions about the history of snakebite in their household. Participants in the key informant interviews will be interviewed to understand how data on snakebite risk can be best presented to support their work.

DETAILED DESCRIPTION:
This study aims to understand whether spatial analysis methods can support the assessment and prediction of geographical variation in snakebite risk.

The investigators will analyse data collected from community and health facility surveys conducted in geographically, ecologically and demographically diverse areas of Kenya and Eswatini. Data sources will comprise existing snakebite incidence data from both countries and prospective data collected through adding snakebite questions to planned health/demographic survey platforms where feasible and conducting a small number of stand-alone cluster-sampled surveys to complement this. Selected households will be invited to complete short questionnaires covering sociodemographic details and snakebite history. Survey data will be compared with health facility data collected in the same locations to assess the value and relative bias of different data sources to snakebite risk assessment. Data will be analysed using geostatistical techniques, and predicted risk will be mapped within and beyond sampled locations where appropriate. Our findings will build knowledge on spatial determinants of snakebite within these countries and support development of a risk mapping methodology for snakebite. Identification of high-risk locations will also support advocacy for resources and guide treatment and prevention activities.

Interviews will also be conducted with key stakeholders in healthcare and research fields in Kenya to help us understand the healthcare decision-making process and how outputs from spatial analysis of snakebite data can be best presented to support this. Interview results will aid development of recommendations for the optimal presentation of snakebite data to support programmatic decision making.

ELIGIBILITY:
Inclusion Criteria:

Household Screening Questionnaire:

* All heads of household from randomly selected households.
* To account for all household members

Snakebite Details Questionnaire:

• All household members with a history of snakebite. If the household member is deceased, a responsible adult from the household will be asked to complete the questionnaire.

Key informant interviews:

* Key informants identified through a stakeholder mapping exercise as having power and/or influence in healthcare decision making or research with relation to Neglected Tropical Diseases/snakebite.
* Willing and motivated to be interviewed

Exclusion Criteria:

Household Screening Questionnaire:

* Households where the household head/a responsible adult is not present at first visit or revisit.
* Household where the household head/responsible adult is unable or unwilling to give consent

Snakebite Details Questionnaire:

• The household member is unable/unwilling to give consent and (in the case of the former) there is no responsible adult available/willing to complete the questionnaire on their behalf

Key informant interviews:

* A participant whose role and organisation has already been represented in the key informant interviews
* Participant declines to be interviewed

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community surveys
  * Populations resident within selected counties.
  Key informant interviews:
  * Those with power and/or influence in healthcare decision making or research with relation to Neglected Tropical Diseases/snakebite.
Sampling Method: Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Geostatistical model of snakebite risk in Kenya and Eswatini | Through study completion, estimated end of 2024
  A geostatistical model of snakebite risk, detailing the statistical association between selected covariates and snakebite risk, based on analysis of data on snakebite incidence collected from contrasting locations in Kenya and Eswatini.
An assessment of the accuracy of snakebite incidence data reported from routine surveillance systems relative to community survey estimates | Through study completion, estimated end of 2024
  An assessment of the accuracy of routine surveillance data sources in relation to community survey incidence estimates (the gold standard measure) in each study location.
Recommendations | Through study completion, estimated end of 2024
  A thematic analysis of key informant interviews on the potential role of and key features needed in snakebite risk maps in order for them to provide utility in healthcare decision making and a set of recommendations to guide presentation of spatial outputs on snakebite risk.

CONTACTS AND LOCATIONS:
Overall Officials: Collinson, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- KSRIC, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Anonymised quantitative datasets (excluding household GPS) and the R code used for analysis will be made available.
Supporting Information: Analytic Code
Time Frame: following study completion and publication of key study outputs